CLINICAL TRIAL: NCT04615988
Title: Correlation of Serum Vitamin D Level with the Development of Endocrine Autoimmune Complications During Treatment with Immune Checkpoint Inhibitors
Brief Title: Correlation Vitamin D Level to Endocrine Autoimmune Toxicity Due to Immune Checkpoint Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Philip Friedlander, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 19-1977
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Thyroid; PD-1; Cancer
Keywords: vitamin D deficiency; immunotherapy with inhibitor of PD-1/L1; immune mediated thyroid toxicity
MeSH Terms: conditions — Thyroid Diseases; Neoplasms; Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants being treated with immunotherapy: Participants who are to receive standard of care immunotherapy targeting PD-1 or PDL1 as treatment for malignancy
  Interventions: Other: blood draw and questionnaire completion; Other: questionnaire completion, blood collection

INTERVENTIONS:
Other: blood draw and questionnaire completion — questionaires provided to subjects during visits while on study and baseline one tube of blood drawn
Other: questionnaire completion, blood collection — questionnaire provided to subject during study visits. One tube blood collected for research purposes at baseline

SUMMARY:
The purpose of this research study is to see if the amount of vitamin D in ones blood makes it more or less likely to develop thyroid gland toxicity when being treated with immunotherapy that blocks the activity of proteins called programed death-1(PD-1) or programmed death ligand-1 (PD-L1). Immunotherapy is treatment that makes changes to the immune system to try to fight cancer. Immunotherapy treatments that block the activity of important parts of the immune system called PD-1 and PD-L1 are used to standardly treat many different types of cancer and can cause thyroid toxicity in certain people. In this study the treatment for your cancer is not research treatment but standard of care determined by your oncologist. Blood will be drawn before starting treatment to determine the amount of Vitamin D and also to assess thyroid function. Also questionnaires will be completed before starting treatment and while on treatment to assess symptoms you are experiencing.

DETAILED DESCRIPTION:
Until 2011 no therapy with proven overall survival benefit was Food and Drug Administration (FDA) approved for the treatment of stage IV (disseminated) melanoma. In 2011 ipilimumab, an inhibitor of CTLA-4, was FDA approved for the treatment of stage IV melanoma representing the first immunotherapy to confer an increase in overall survival. CTLA-4 is expressed on the surface of activated T cells and binds to B7 on antigen-presenting cells with higher affinity than the co-stimulatory protein CD28. By competing for and disrupting the binding of CD28 to B7, CTLA-4 prevents T-cell co-stimulation which leads to a dampening of the immune response. Ipilimumab is an IgG1 monoclonal antibody that binds CTLA-4 in an inhibitory manner. Treating stage IV melanoma with ipilimumab confers an overall survival benefit when compared in randomized fashion to peptide vaccine treatment, with median survival increasing from 6 to 10 months and 2-year survival increasing from 14% to 24%. Benefit is durable as the overall survival rate plateauing at 21% by year 3 with follow-up extending up to 10 years.

The regulation of immune T-cell activity is complex involving multiple activating and inhibitory protein interactions with antigen presenting cells. T-cells express the protein programmed death-1 (PD-1) which when bound to its ligand PD-L1 normally expressed on peripheral tissues inhibits T-cell activity. Many melanomas select for aberrant expression of PD-L1. When T-cells infiltrate the melanoma metastasis tumor microenvironment the PD-1 on the infiltrating T-cells binds the tumor expressed PD-L1 leading to inhibition of T-cell activity. Blocking the interaction of PD-1 to PD-L1 in stage IV melanoma leads to clinical efficacy. Two inhibitors of PD-1, nivolumab and pembrolizumab, were FDA approved in 2014 for the treatment stage IV melanoma with response rates approximating 40% and 5-year survival post-nivolumab treatment of 35%. In 2015 concurrent treatment with ipilimumab and nivolumab was FDA-approved on the basis of a 57.6% response rate.

Ipilimumab is infused intravenously as a single agent every 3 weeks for a total of four treatments. Nivolumab is administered intravenously every two weeks at dose of 240 mg or every four weeks at a dose of 480 mg while pembrolizumab is infused every three weeks at dose of 200 mg or every 6 weeks at 400 mg per dose. With concurrent ipilimumab and nivolumab treatment the combination is administered every three weeks for 4 doses and then nivolumab is infused as a single agent every two weeks.

The inhibition of immune cell activity in the tumor microenvironment through the selection of PD-L1 expression on tumor cells is not specific to melanoma. Clinical efficacy has been appreciated in a range of malignancies leading to multiple FDA approvals for stage IV disease. Specifically pembrolizumab is also FDA approved for treatment of stage IV non-small cell lung cancer and recurrent or metastatic HNSCC. Nivolumab is also FDA approved for the treatment of metastatic non-small cell lung cancer, advanced renal cell carcinoma, classical Hodgkin lymphoma, and recurrent or metastatic squamous cell carcinoma of the head and neck.

Given the mechanism of action of CTLA-4 and PD-1 inhibitors toxicity is largely immune mediated. The incidence of grade3 or higher immune mediated toxicity following single agent ipilimumab treatment is approximately 25%. Following nivolumab or pembrolizumab treatment the risk of such toxicity is 17-20% while following combined ipilimumab and nivolumab treatment the risk is 55-59%. Toxicity can manifest based on organ or tissue involved such as rash, colitis, hepatitis, nephritis, pancreatitis, myocarditis, pneumonitis uveitis, neurologic or endocrine.

Autoimmune endocrinopathies (thyroid disease, hypophysitis, adrenal failure and diabetes) have been reported in 6-25% of patients on anti-PD-1 therapies in different case series. With concurrent CTLA-4 and PD-1 inhibition the rate of thyroid immune mediated toxicity is approximately 15%. Autoimmune thyroid disease can easily be detected on routine blood tests before the patient develops symptoms, is associated with known autoantibodies that have clinical assays, and autoimmune thyroid disease can be treated with thyroid hormone replacement, if needed.

Serum 25-hydroxyvitamin D levels have been inversely correlated with the levels of anti-thyroperoxidase (TPO) antibodies in some cohorts. Vitamin D deficiency has also been linked to an increased risk of autoimmune thyroid disease. Vitamin D supplementation has been reported to suppress CD4+ T cell and NK cell function in pre-clinical and clinical studies. It is not known whether vitamin D deficiency plays a role in the development of the irAEs in patients treated with immune checkpoint inhibitors. Furthermore, it is not known if vitamin D deficiency or supplementation alters the rate of response to immune checkpoint inhibitors.

PD-1/PD-L1 inhibition has demonstrated clinical efficacy in a range of malignancies with treatment leading to durable benefit. However this type of treatment can lead to immune mediated toxicity that if high grade can necessitate interventions or management with high dose steroids. As such identifying biomarkers for toxicity and strategies to minimize toxicity risk are very important. Serum 25-hydroxyvitamin D levels have been inversely correlated with the levels of anti-thyroperoxidase (TPO) antibodies in some cohorts. Vitamin D deficiency has also been linked to an increased risk of autoimmune thyroid disease. This study plans to determine if baseline deficiency in serum 25-hydroxy vitamin D levels correlates with altered risk of developing immune mediated toxicity of the thyroid gland in patients being treated with anti-PD1/PD-L1 immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Malignancy which the treating oncologist plans for next treatment to inhibit PD-1or PD-L1 with the immune inhibitor being the only immunotherapy. Twenty-five subjects in a separate cohort will need for eligibility to be planned for treatment with anti-PD1/PD-L1 plus antri-CTLA-4 therapy.
* Willingness to complete symptom questionnaires
* Willingness to allow blood draws
* Ability to provide informed consent
* Age > 18 years old

Exclusion Criteria:

* History of clinical or subclinical hyperthyroidism or hypothyroidism
* Hemoglobin < 9
* Inability to come for all study visits.
* Actively on vitamin D supplementation due to vitamin D deficiency (As part of a multivitamin is not exclusionary)
* Pregnant or lactating
* History of hypophysitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are adults age 18 or older with advanced cancer and are planned to receive standard of care treatment with a PD-1/L-1 inhibitor or with standard of care anti-CTLA-4 plus antiPD-1/L1 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with risk of developing autoimmune thyroid disease treated with single agent. | 20 weeks
  Number of participants with risk of developing autoimmune thyroid disease in cancer treated with single agent anti-PD-1/PD-L1 therapy with baseline pre-treatment vitamin D deficiency compared with those with normal vitamin D levels

SECONDARY OUTCOMES:
Number of participants with risk of developing autoimmune thyroid disease treated with two agents. | 20 weeks
  Number of participants with risk of developing autoimmune thyroid disease in cancer patients treated with anti-CTLA-4 + anti-PD-1/PD-L1 therapy in patients with vitamin D deficiency, compared with those with normal vitamin D levels.
Correlation of development high grade immune toxicity from PD-1/PD-L1 inhibitor with baseline vitamin D status (deficient or not) | 20 weeks
  The risk of developing a high grade (> gd 3) immune mediated toxicity in the 20 weeks. following initiation of treatment with a PD-1/PD-L1 inhibitor in cancer patients with baseline vitamin D deficiency will be compared to the risk in those with baseline normal vitamin D levels. Correlate baseline vitamin D status with development of thyroid toxicity.
Baseline Assessment Questionnaire | 20 weeks
  Participants using the Baseline Assessment Questionnaire rate symptoms on scale of 1-10 with higher number reflecting more severe symptom.
On Treatment Symptom Questionnaire | 20 weeks
  Symptom questionnaire using the On Treatment Symptom Questionnaire - full score 1-10 with increasing number reflecting more severe symptom.
Change in Thyroid antibody | baseline and 20 weeks
  Correlate changes in thyroid antibody expression in patients who develop thyroid toxicity and correlation with vitamin D level (low versus normal/high). Thyroid antibody blood tests assessed pre-treatment and rechecked if develop thyroid toxicity and positivity of antibodies compared at the two timepoints.
Correlation vitamin D baseline level to physician assessment of anti-PD-1/L1 | 24 weeks
  Correlate presence or absence of baseline vitamin D deficiency with efficacy of PD-1/PD-L1 immunotherapy based on treating physician's assessment of response or stabilization of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Friedlander, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital /Tisch Cancer Cancer/Ruttenberg Treatment Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No